CLINICAL TRIAL: NCT01584544
Title: Phase I Study of Preoperative Concurrent Chemo-radiation With Capecitabine in Elderly Rectal Cancer Patients
Brief Title: Safety Study of Capecitabine With Radiation in Elderly Rectal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Jing Jin, M.D., vice chair of radiation department, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CH-GI-024
Record Dates: First submitted 2012-04-20; First posted 2012-04-25 (Estimated); Results first posted 2015-04-20 (Estimated); Last update posted 2015-04-20 (Estimated); Status verified 2015-04

CONDITIONS: Rectal Neoplasms
Keywords: rectal neoplasms; aged; chemoradiotherapy; clinical trials, phase I; capecitabine
MeSH Terms: conditions — Rectal Neoplasms | interventions — Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- 1000mg (Experimental): capecitabine 1000mg/m2/d d1-14, d22-25 combined with concurrent radiotherapy will be given to enrolled patients.
  Interventions: Drug: capecitabine
- 1200mg (Experimental): capecitabine 1200mg/m2/d d1-14, d22-35 combined with concurrent radiotherapy will be given to enrolled patients.
  Interventions: Drug: Capecitabine
- 1350mg (Experimental): capecitabine 1300mg/m2/d d1-14, d22-35 combined with concurrent radiotherapy will be given to enrolled patients.
  Interventions: Drug: Capecitabine
- 1500mg (Experimental): capecitabine 1500mg/m2/d d1-14, d22-35 combined with concurrent radiotherapy will be given to enrolled patients.
  Interventions: Drug: Capecitabine
- 1650mg (Experimental): capecitabine 1650mg/m2/d d1-14, d22-35 combined with concurrent radiotherapy will be given to enrolled patients.
  Interventions: Drug: Capecitabine

INTERVENTIONS:
Drug: capecitabine — oral pills, 1000mg/m2/d, split in two times, d1-14, d22-35 combined with concurrent pelvic radiation
  Other Names: stare 1
  Arms: 1000mg
Drug: Capecitabine — oral pills, 1200mg/m2/d, split in two times, d1-14, d22-35 combined with concurrent pelvic radiation
  Other Names: stare 2
  Arms: 1200mg
Drug: Capecitabine — oral pills, 1350mg/m2/d, split in two times, d1-14, d22-35 combined with concurrent pelvic radiation
  Other Names: stare 3
  Arms: 1350mg
Drug: Capecitabine — oral pills, 1500mg/m2/d, split in two times, d1-14, d22-35 combined with concurrent pelvic radiation
  Other Names: stare 4
  Arms: 1500mg
Drug: Capecitabine — oral pills, 1650mg/m2/d, split in two times, d1-14, d22-35 combined with concurrent pelvic radiation
  Other Names: stare 5
  Arms: 1650mg

SUMMARY:
This phase I study is designed to determine the maximum tolerant dose of capecitabine when used in preoperative concurrent chemo-radiation for locally advanced rectal patients over 75 years old.

DETAILED DESCRIPTION:
It is proved that preoperative concurrent chemo-radiotherapy can improve both local control and overall survival in stage II/III rectal cancer patients. But elderly patients, especially patients over 75 years were hardly involved in related clinical trials considered of their fragility.

Several retrospective study showed that old rectal cancer patients would also benefit from concurrent chemo-radiation, with acceptable toxicity. Several new drug, such as capecitabine, also seem to be safety for elderly cancer patients. But few prospective study has been carried out.

The investigators designed this phase I study, to explore the maximum tolerant dose of capecitabine in preoperative concurrent chemoradiation for elderly stage II/III rectal cancer patients, as well as to evaluate safety.

ELIGIBILITY:
Inclusion Criteria:

* rectal adenocarcinoma, clinical stage II/III(T3-4 or N+, AJCC 7th).
* KPS status no less than 70; Charlson comorbidity no more than 3.
* life expectancy more than 6 months.
* hemoglobin >= 100g/L, white blood cell >= 3.5*10E9/L, neutrophil >= 1.5*10E9/L, platelet >= 100*10E9/L.Creatin normal, Total bilirubin normal, AST and AST normal, AKP normal.
* do not have allergy history to thymidine phosphorylase.
* do not receive surgery ( except palliative colostomy) or chemotherapy or other anti-cancer treatment
* no previously pelvic irradiation history
* informed consent signed

Exclusion Criteria:

* other cancer history, except curable non-melanoma skin cancer or cervix in-situ carcinoma
* previous pelvic irradiation history
* receiving surgery (except palliative colostomy), chemotherapy or other anti-cancer treatment
* allergy history to thymidine phosphorylase
* active infection existed
* severe complication, such as acute myocardial infarction in 6 months, uncontrolled diabetes ( Plasma glucose concentrations in any time of a day≥11.1mmol/L）, severe cardiac arrhythmia， etc.
* anticipate other clinical trials in four weeks before enrollment

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 24 (Actual)
Dates: Start 2011-01; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jing Jin, Ph.D., Principal Investigator — Chinese Academic Medical Science; Yexiong Li, Ph.D., Principal Investigator — Chinese Academic Medical Science
Locations (1):
- radiation department, Cancer Hospital, CAMS, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Aapro MS, Kohne CH, Cohen HJ, Extermann M. Never too old? Age should not be a barrier to enrollment in cancer clinical trials. Oncologist. 2005 Mar;10(3):198-204. doi: 10.1634/theoncologist.10-3-198. PMID 15793223
- [Background] Papamichael D, Audisio R, Horiot JC, Glimelius B, Sastre J, Mitry E, Van Cutsem E, Gosney M, Kohne CH, Aapro M; SIOG. Treatment of the elderly colorectal cancer patient: SIOG expert recommendations. Ann Oncol. 2009 Jan;20(1):5-16. doi: 10.1093/annonc/mdn532. Epub 2008 Oct 15. PMID 18922882
- [Background] Potosky AL, Harlan LC, Kaplan RS, Johnson KA, Lynch CF. Age, sex, and racial differences in the use of standard adjuvant therapy for colorectal cancer. J Clin Oncol. 2002 Mar 1;20(5):1192-202. doi: 10.1200/JCO.2002.20.5.1192. PMID 11870160
- [Background] Hemminki K, Santi I, Weires M, Thomsen H, Sundquist J, Bermejo JL. Tumor location and patient characteristics of colon and rectal adenocarcinomas in relation to survival and TNM classes. BMC Cancer. 2010 Dec 21;10:688. doi: 10.1186/1471-2407-10-688. PMID 21176147
- [Background] Janssen-Heijnen ML, Houterman S, Lemmens VE, Louwman MW, Maas HA, Coebergh JW. Prognostic impact of increasing age and co-morbidity in cancer patients: a population-based approach. Crit Rev Oncol Hematol. 2005 Sep;55(3):231-40. doi: 10.1016/j.critrevonc.2005.04.008. PMID 15979890
- [Background] Chang GJ, Skibber JM, Feig BW, Rodriguez-Bigas M. Are we undertreating rectal cancer in the elderly? An epidemiologic study. Ann Surg. 2007 Aug;246(2):215-21. doi: 10.1097/SLA.0b013e318070838f. PMID 17667499
- [Background] Townsley C, Pond GR, Peloza B, Kok J, Naidoo K, Dale D, Herbert C, Holowaty E, Straus S, Siu LL. Analysis of treatment practices for elderly cancer patients in Ontario, Canada. J Clin Oncol. 2005 Jun 1;23(16):3802-10. doi: 10.1200/JCO.2005.06.742. PMID 15923574
- [Background] Ayanian JZ, Zaslavsky AM, Fuchs CS, Guadagnoli E, Creech CM, Cress RD, O'Connor LC, West DW, Allen ME, Wolf RE, Wright WE. Use of adjuvant chemotherapy and radiation therapy for colorectal cancer in a population-based cohort. J Clin Oncol. 2003 Apr 1;21(7):1293-300. doi: 10.1200/JCO.2003.06.178. PMID 12663717
- [Background] Surgery for colorectal cancer in elderly patients: a systematic review. Colorectal Cancer Collaborative Group. Lancet. 2000 Sep 16;356(9234):968-74. PMID 11041397
- [Background] Vulto AJ, Lemmens VE, Louwman MW, Janssen-Heijnen ML, Poortmans PH, Lybeert ML, Coebergh JW. The influence of age and comorbidity on receiving radiotherapy as part of primary treatment for cancer in South Netherlands, 1995 to 2002. Cancer. 2006 Jun 15;106(12):2734-42. doi: 10.1002/cncr.21934. PMID 16703598
- [Background] Devon KM, Vergara-Fernandez O, Victor JC, McLeod RS. Colorectal cancer surgery in elderly patients: presentation, treatment, and outcomes. Dis Colon Rectum. 2009 Jul;52(7):1272-7. doi: 10.1007/DCR.0b013e3181a74d2e. PMID 19571704
- [Background] Law WL, Choi HK, Ho JW, Lee YM, Seto CL. Outcomes of surgery for mid and distal rectal cancer in the elderly. World J Surg. 2006 Apr;30(4):598-604. doi: 10.1007/s00268-005-0442-x. PMID 16568224
- [Background] Endreseth BH, Romundstad P, Myrvold HE, Bjerkeset T, Wibe A; Norwegian Rectal Cancer Group. Rectal cancer treatment of the elderly. Colorectal Dis. 2006 Jul;8(6):471-9. doi: 10.1111/j.1463-1318.2005.00921.x. PMID 16784465
- [Background] Larsen SG, Wiig JN, Tretli S, Giercksky KE. Surgery and pre-operative irradiation for locally advanced or recurrent rectal cancer in patients over 75 years of age. Colorectal Dis. 2006 Mar;8(3):177-85. doi: 10.1111/j.1463-1318.2005.00877.x. PMID 16466556
- [Background] Vironen JH, Sainio P, Husa AI, Kellokumpu IH. Complications and survival after surgery for rectal cancer in patients younger than and aged 75 years or older. Dis Colon Rectum. 2004 Jul;47(7):1225-31. doi: 10.1007/s10350-004-0557-4. Epub 2004 May 28. PMID 15164247
- [Background] Barrier A, Ferro L, Houry S, Lacaine F, Huguier M. Rectal cancer surgery in patients more than 80 years of age. Am J Surg. 2003 Jan;185(1):54-7. doi: 10.1016/s0002-9610(02)01120-0. PMID 12531446
- [Background] Rutten H, den Dulk M, Lemmens V, Nieuwenhuijzen G, Krijnen P, Jansen-Landheer M, van de Poll Franse L, Coebergh JW, Martijn H, Marijnen C, van de Velde C. Survival of elderly rectal cancer patients not improved: analysis of population based data on the impact of TME surgery. Eur J Cancer. 2007 Oct;43(15):2295-300. doi: 10.1016/j.ejca.2007.07.009. Epub 2007 Aug 20. PMID 17709242
- [Background] Rutten HJ, den Dulk M, Lemmens VE, van de Velde CJ, Marijnen CA. Controversies of total mesorectal excision for rectal cancer in elderly patients. Lancet Oncol. 2008 May;9(5):494-501. doi: 10.1016/S1470-2045(08)70129-3. PMID 18452860
- [Background] Sargent DJ, Goldberg RM, Jacobson SD, Macdonald JS, Labianca R, Haller DG, Shepherd LE, Seitz JF, Francini G. A pooled analysis of adjuvant chemotherapy for resected colon cancer in elderly patients. N Engl J Med. 2001 Oct 11;345(15):1091-7. doi: 10.1056/NEJMoa010957. PMID 11596588
- [Background] Iwashyna TJ, Lamont EB. Effectiveness of adjuvant fluorouracil in clinical practice: a population-based cohort study of elderly patients with stage III colon cancer. J Clin Oncol. 2002 Oct 1;20(19):3992-8. doi: 10.1200/JCO.2002.03.083. PMID 12351596
- [Background] Sundararajan V, Mitra N, Jacobson JS, Grann VR, Heitjan DF, Neugut AI. Survival associated with 5-fluorouracil-based adjuvant chemotherapy among elderly patients with node-positive colon cancer. Ann Intern Med. 2002 Mar 5;136(5):349-57. doi: 10.7326/0003-4819-136-5-200203050-00007. PMID 11874307
- [Background] Goldberg RM, Tabah-Fisch I, Bleiberg H, de Gramont A, Tournigand C, Andre T, Rothenberg ML, Green E, Sargent DJ. Pooled analysis of safety and efficacy of oxaliplatin plus fluorouracil/leucovorin administered bimonthly in elderly patients with colorectal cancer. J Clin Oncol. 2006 Sep 1;24(25):4085-91. doi: 10.1200/JCO.2006.06.9039. PMID 16943526
- [Background] Pignon T, Horiot JC, Bolla M, van Poppel H, Bartelink H, Roelofsen F, Pene F, Gerard A, Einhorn N, Nguyen TD, Vanglabbeke M, Scalliet P. Age is not a limiting factor for radical radiotherapy in pelvic malignancies. Radiother Oncol. 1997 Feb;42(2):107-20. doi: 10.1016/s0167-8140(96)01861-0. PMID 9106920
- [Background] Preoperative short-term radiation therapy in operable rectal carcinoma. A prospective randomized trial. Stockholm Rectal Cancer Study Group. Cancer. 1990 Jul 1;66(1):49-55. doi: 10.1002/1097-0142(19900701)66:13.0.co;2-1. PMID 2191763
- [Background] Holm T, Rutqvist LE, Johansson H, Cedermark B. Postoperative mortality in rectal cancer treated with or without preoperative radiotherapy: causes and risk factors. Br J Surg. 1996 Jul;83(7):964-8. doi: 10.1002/bjs.1800830725. PMID 8813788
- [Background] Randomized study on preoperative radiotherapy in rectal carcinoma. Stockholm Colorectal Cancer Study Group. Ann Surg Oncol. 1996 Sep;3(5):423-30. doi: 10.1007/BF02305759. PMID 8876883
- [Background] Shahir MA, Lemmens VE, van de Poll-Franse LV, Voogd AC, Martijn H, Janssen-Heijnen ML. Elderly patients with rectal cancer have a higher risk of treatment-related complications and a poorer prognosis than younger patients: a population-based study. Eur J Cancer. 2006 Nov;42(17):3015-21. doi: 10.1016/j.ejca.2005.10.032. Epub 2006 Jun 22. PMID 16797967
- [Background] Lorchel F, Peignaux K, Crehange G, Bosset M, Puyraveau M, Mercier M, Bosset JF, Maingon P. Preoperative radiotherapy in elderly patients with rectal cancer. Gastroenterol Clin Biol. 2007 Apr;31(4):436-41. doi: 10.1016/s0399-8320(07)89407-3. PMID 17483785
- [Background] Fiorica F, Cartei F, Carau B, Berretta S, Sparta D, Tirelli U, Santangelo A, Maugeri D, Luca S, Leotta C, Sorace R, Berretta M. Adjuvant radiotherapy on older and oldest elderly rectal cancer patients. Arch Gerontol Geriatr. 2009 Jul-Aug;49(1):54-9. doi: 10.1016/j.archger.2008.05.001. Epub 2008 Jun 24. PMID 18573548
- [Background] Pasetto LM, Basso U, Friso ML, Pucciarelli S, Agostini M, Rugge M, Sinigaglia G, Lise M, Sotti G, Monfardini S. Determining therapeutic approaches in the elderly with rectal cancer. Drugs Aging. 2007;24(9):781-90. doi: 10.2165/00002512-200724090-00006. PMID 17727307
- [Background] Neugut AI, Fleischauer AT, Sundararajan V, Mitra N, Heitjan DF, Jacobson JS, Grann VR. Use of adjuvant chemotherapy and radiation therapy for rectal cancer among the elderly: a population-based study. J Clin Oncol. 2002 Jun 1;20(11):2643-50. doi: 10.1200/JCO.2002.08.062. PMID 12039925
- [Background] Dobie SA, Warren JL, Matthews B, Schwartz D, Baldwin LM, Billingsley K. Survival benefits and trends in use of adjuvant therapy among elderly stage II and III rectal cancer patients in the general population. Cancer. 2008 Feb 15;112(4):789-99. doi: 10.1002/cncr.23244. PMID 18189291
- [Background] Pasetto LM, Friso ML, Pucciarelli S, Basso U, Falci C, Bortolami A, Toppan P, Agostini M, Rugge M, Serpentini S, Nitti D, Monfardini S. Rectal cancer neoadjuvant treatment in elderly patients. Anticancer Res. 2006 Sep-Oct;26(5B):3913-23. PMID 17094422
- [Background] Hutchins LF, Unger JM, Crowley JJ, Coltman CA Jr, Albain KS. Underrepresentation of patients 65 years of age or older in cancer-treatment trials. N Engl J Med. 1999 Dec 30;341(27):2061-7. doi: 10.1056/NEJM199912303412706. PMID 10615079
- [Background] Lewis JH, Kilgore ML, Goldman DP, Trimble EL, Kaplan R, Montello MJ, Housman MG, Escarce JJ. Participation of patients 65 years of age or older in cancer clinical trials. J Clin Oncol. 2003 Apr 1;21(7):1383-9. doi: 10.1200/JCO.2003.08.010. PMID 12663731
- [Background] Ceelen W, Fierens K, Van Nieuwenhove Y, Pattyn P. Preoperative chemoradiation versus radiation alone for stage II and III resectable rectal cancer: a systematic review and meta-analysis. Int J Cancer. 2009 Jun 15;124(12):2966-72. doi: 10.1002/ijc.24247. PMID 19253365
- [Background] Fiorica F, Cartei F, Licata A, Enea M, Ursino S, Colosimo C, Camma C. Can chemotherapy concomitantly delivered with radiotherapy improve survival of patients with resectable rectal cancer? A meta-analysis of literature data. Cancer Treat Rev. 2010 Nov;36(7):539-49. doi: 10.1016/j.ctrv.2010.03.002. Epub 2010 Mar 23. PMID 20334979
- [Background] Sauer R, Becker H, Hohenberger W, Rodel C, Wittekind C, Fietkau R, Martus P, Tschmelitsch J, Hager E, Hess CF, Karstens JH, Liersch T, Schmidberger H, Raab R; German Rectal Cancer Study Group. Preoperative versus postoperative chemoradiotherapy for rectal cancer. N Engl J Med. 2004 Oct 21;351(17):1731-40. doi: 10.1056/NEJMoa040694. PMID 15496622
- [Background] Bujko K, Kepka L, Michalski W, Nowacki MP. Does rectal cancer shrinkage induced by preoperative radio(chemo)therapy increase the likelihood of anterior resection? A systematic review of randomised trials. Radiother Oncol. 2006 Jul;80(1):4-12. doi: 10.1016/j.radonc.2006.04.012. Epub 2006 May 26. PMID 16730086
- [Background] Wong RK, Tandan V, De Silva S, Figueredo A. Pre-operative radiotherapy and curative surgery for the management of localized rectal carcinoma. Cochrane Database Syst Rev. 2007 Apr 18;(2):CD002102. doi: 10.1002/14651858.CD002102.pub2. PMID 17443515
- [Background] Roels S, Duthoy W, Haustermans K, Penninckx F, Vandecaveye V, Boterberg T, De Neve W. Definition and delineation of the clinical target volume for rectal cancer. Int J Radiat Oncol Biol Phys. 2006 Jul 15;65(4):1129-42. doi: 10.1016/j.ijrobp.2006.02.050. Epub 2006 Jun 5. PMID 16750329
- [Background] Tepper JE, O'Connell M, Niedzwiecki D, Hollis DR, Benson AB 3rd, Cummings B, Gunderson LL, Macdonald JS, Martenson JA, Mayer RJ. Adjuvant therapy in rectal cancer: analysis of stage, sex, and local control--final report of intergroup 0114. J Clin Oncol. 2002 Apr 1;20(7):1744-50. doi: 10.1200/JCO.2002.07.132. PMID 11919230
- [Background] O'Connell MJ, Martenson JA, Wieand HS, Krook JE, Macdonald JS, Haller DG, Mayer RJ, Gunderson LL, Rich TA. Improving adjuvant therapy for rectal cancer by combining protracted-infusion fluorouracil with radiation therapy after curative surgery. N Engl J Med. 1994 Aug 25;331(8):502-7. doi: 10.1056/NEJM199408253310803. PMID 8041415
- [Background] Van Cutsem E, Twelves C, Cassidy J, Allman D, Bajetta E, Boyer M, Bugat R, Findlay M, Frings S, Jahn M, McKendrick J, Osterwalder B, Perez-Manga G, Rosso R, Rougier P, Schmiegel WH, Seitz JF, Thompson P, Vieitez JM, Weitzel C, Harper P; Xeloda Colorectal Cancer Study Group. Oral capecitabine compared with intravenous fluorouracil plus leucovorin in patients with metastatic colorectal cancer: results of a large phase III study. J Clin Oncol. 2001 Nov 1;19(21):4097-106. doi: 10.1200/JCO.2001.19.21.4097. PMID 11689577
- [Background] Hoff PM, Ansari R, Batist G, Cox J, Kocha W, Kuperminc M, Maroun J, Walde D, Weaver C, Harrison E, Burger HU, Osterwalder B, Wong AO, Wong R. Comparison of oral capecitabine versus intravenous fluorouracil plus leucovorin as first-line treatment in 605 patients with metastatic colorectal cancer: results of a randomized phase III study. J Clin Oncol. 2001 Apr 15;19(8):2282-92. doi: 10.1200/JCO.2001.19.8.2282. PMID 11304782
- [Background] Twelves C; Xeloda Colorectal Cancer Group. Capecitabine as first-line treatment in colorectal cancer. Pooled data from two large, phase III trials. Eur J Cancer. 2002 Feb;38 Suppl 2:15-20. doi: 10.1016/s0959-8049(01)00415-4. PMID 11841931
- [Background] Twelves C, Wong A, Nowacki MP, Abt M, Burris H 3rd, Carrato A, Cassidy J, Cervantes A, Fagerberg J, Georgoulias V, Husseini F, Jodrell D, Koralewski P, Kroning H, Maroun J, Marschner N, McKendrick J, Pawlicki M, Rosso R, Schuller J, Seitz JF, Stabuc B, Tujakowski J, Van Hazel G, Zaluski J, Scheithauer W. Capecitabine as adjuvant treatment for stage III colon cancer. N Engl J Med. 2005 Jun 30;352(26):2696-704. doi: 10.1056/NEJMoa043116. PMID 15987918
- [Background] Dunst J, Reese T, Sutter T, Zuhlke H, Hinke A, Kolling-Schlebusch K, Frings S. Phase I trial evaluating the concurrent combination of radiotherapy and capecitabine in rectal cancer. J Clin Oncol. 2002 Oct 1;20(19):3983-91. doi: 10.1200/JCO.2002.02.049. PMID 12351595
- [Background] Ngan SY, Michael M, Mackay J, McKendrick J, Leong T, Lim Joon D, Zalcberg JR. A phase I trial of preoperative radiotherapy and capecitabine for locally advanced, potentially resectable rectal cancer. Br J Cancer. 2004 Sep 13;91(6):1019-24. doi: 10.1038/sj.bjc.6602106. PMID 15305186
- [Background] Jin J, Li YX, Liu YP, Wang WH, Song YW, Li T, Li N, Yu ZH, Liu XF. A phase I study of concurrent radiotherapy and capecitabine as adjuvant treatment for operable rectal cancer. Int J Radiat Oncol Biol Phys. 2006 Mar 1;64(3):725-9. doi: 10.1016/j.ijrobp.2005.08.017. Epub 2005 Oct 19. PMID 16242260
- [Background] Kim DY, Jung KH, Kim TH, Kim DW, Chang HJ, Jeong JY, Kim YH, Son SH, Yun T, Hong CW, Sohn DK, Lim SB, Choi HS, Jeong SY, Park JG. Comparison of 5-fluorouracil/leucovorin and capecitabine in preoperative chemoradiotherapy for locally advanced rectal cancer. Int J Radiat Oncol Biol Phys. 2007 Feb 1;67(2):378-84. doi: 10.1016/j.ijrobp.2006.08.063. Epub 2006 Nov 9. PMID 17097835
- [Background] Ramani VS, Sun Myint A, Montazeri A, Wong H. Preoperative chemoradiotherapy for rectal cancer: a comparison between intravenous 5-fluorouracil and oral capecitabine. Colorectal Dis. 2010 Aug;12 Suppl 2:37-46. doi: 10.1111/j.1463-1318.2010.02323.x. PMID 20618366
- [Background] Feliu J, Escudero P, Llosa F, Bolanos M, Vicent JM, Yubero A, Sanz-Lacalle JJ, Lopez R, Lopez-Gomez L, Casado E, Gomez-Reina MJ, Gonzalez-Baron M. Capecitabine as first-line treatment for patients older than 70 years with metastatic colorectal cancer: an oncopaz cooperative group study. J Clin Oncol. 2005 May 1;23(13):3104-11. doi: 10.1200/JCO.2005.06.035. PMID 15860870
- [Background] Pasetto LM, Monfardini S. The role of capecitabine in the treatment of colorectal cancer in the elderly. Anticancer Res. 2006 May-Jun;26(3B):2381-6. PMID 16821620

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 1000mg | 1200mg | 1350mg | 1500mg | 1650mg
Started | 3 | 6 | 6 | 3 | 6
Completed | 3 | 6 | 6 | 3 | 6
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1000mg | 1200mg | 1350mg | 1500mg | 1650mg | Total
Number analyzed (Participants) | 3 | 6 | 6 | 3 | 6 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0 | 0
  >=65 years | 3 | 6 | 6 | 3 | 6 | 24
Age, Continuous [Median (Full Range); unit: years] | 77 [75 to 82] | 77 [75 to 84] | 78 [75 to 82] | 76 [76 to 77] | 78 [76 to 79] | 78 [75 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 2 | 1 | 4 | 11
  Male | 2 | 3 | 4 | 2 | 2 | 13
Region of Enrollment [Number; unit: participants]
  China | 3 | 6 | 6 | 3 | 6 | 24

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experienced Dose Limited Toxicity
Description: Dose related toxicity is defined as follows:1. luecopenia > grade 2; granular cell decrease > grade 2; anemia > grade 1; platelet > grade 1;SGPT/SGOT elevation > grade 1; ALP > grade 1; GGT > grade 1; Tbil > grade 1;renal function damag > grade 2;Non-gradular cell decreased fever > grade 1;nausea/vomiting > grade 1; fatigue > grade 2; weight loss > grade 2;gastritis > grade 2; dairrea > grade 2; abdominal pain > grade 2; upper gastrointestinal bleeding > grade 1;other toxic reaction > grade 2;KPS < 50 during the treatment
Time Frame: up to 7 weeks from start of the treatment
Measure: Number; unit: participants
Arm/Group | 1000mg | 1200mg | 1350mg | 1500mg | 1650mg
Number analyzed (Participants) | 3 | 6 | 6 | 3 | 6
participants | 0 | 1 | 1 | 0 | 1

ADVERSE EVENTS:
Time Frame: 7 weeks after treatment started
Arm/Group | 1000mg | 1200mg | 1350mg | 1500mg | 1650mg
Serious Adverse Events (participants affected / at risk) | 0/3 | 1/6 | 1/6 | 0/3 | 1/6
Other Adverse Events (participants affected / at risk) | 3/3 | 6/6 | 6/6 | 3/3 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 1000mg (N=3) | 1200mg (N=6) | 1350mg (N=6) | 1500mg (N=3) | 1650mg (N=6)
Diarrhea, Grade 3 (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Lung infection, Grade 3 (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Proctitis, Grade 3 (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Fever, Grade 3 (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Fatigue, Grade 3 (General disorders) | 0 | 0 | 0 | 0 | 1
Pain, Grade 3 (General disorders) | 0 | 0 | 0 | 0 | 1
Nausea, Grade 3 (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 1000mg (N=3) | 1200mg (N=6) | 1350mg (N=6) | 1500mg (N=3) | 1650mg (N=6)
Radiation dermatitis (Skin and subcutaneous tissue disorders) | 3 | 6 | 5 | 3 | 2
Diarrhea (Gastrointestinal disorders) | 1 | 5 | 1 | 1 | 3
Fatigue (General disorders) | 2 | 1 | 2 | 2 | 2
Pain (General disorders) | 0 | 3 | 2 | 1 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 3 | 2 | 3
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 3
Proctitis (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0
Fever (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 2 | 4 | 5 | 2 | 2
Anemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Hand-foot syndrome (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Weight loss (General disorders) | 0 | 0 | 1 | 0 | 0
Urinary frequency (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No